CLINICAL TRIAL: NCT06603051
Title: The Effect of Pre-Operative Cryoneurolysis on Post-Operative Narcotic Consumption in Patients Undergoing Autograft ACL Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virtua Health, Inc. (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G24064; CON-000367 (Other Grant/Funding Number: Pacira Bioscience Inc.)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: ACL Repair
Keywords: ACL Repair; Cryoneurolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A: ACL reconstruction usual care (No Intervention): On the day of surgery, all patients (Group A and Group B) will receive a multi-modal oral pre-operative cocktail and an ultrasound guided adductor canal block. Additionally, an ultrasound guided popliteal or infiltration of the tissue plane between the popliteal artery and the capsule of the knee (iPACK) block will be administered. The pre-operative oral medication cocktail and block medications are as follows: Acetaminophen 975 mg x 1, Celecoxib 400 mg PO x 1, adductor canal block with 133 mg (10 mL) liposomal bupivacaine (EXPAREL) admixed with 0.5% bupivacaine HCl 50 mg (10 mL), popliteal or iPACK nerve infiltration with 133 mg (10 mL) liposomal bupivacaine (EXPAREL) admixed with 0.5% bupivacaine HCl 50 mg (10 mL). 15 mg IV ketorolac at conclusion of the case will be administered.
- Arm B: Usual care plus pre-operative cryoneurolysis (Experimental): Those randomized to the intervention group (Group B) will receive a standard treatment of Cryoneurolysis to their surgical knee within 7-10 days of their scheduled surgery. Treatment nerves for the procedure will include the anterior femoral cutaneous nerve (AFCN), supra-patellar branch of the saphenous nerve (SPBSN) and infra-patellar branch of the saphenous nerve (IPBSN).
  Interventions: Procedure: Cryoneurolysis

INTERVENTIONS:
Procedure: Cryoneurolysis — Those randomized to the intervention group (Group B) will receive a standard treatment of Cryoneurolysis to their surgical knee within 7-10 days of their scheduled surgery. Treatment nerves for the procedure will include the anterior femoral cutaneous nerve (AFCN), supra-patellar branch of the saphenous nerve (SPBSN) and infra-patellar branch of the saphenous nerve (IPBSN).
  Arms: Arm B: Usual care plus pre-operative cryoneurolysis

SUMMARY:
The purpose of the research is to investigate the effect of preoperative Cryoneurolysis of the knee on postoperative pain management in patients undergoing autograft anterior cruciate ligament (ACL) reconstruction (a surgical procedure that makes a new ACL using the patient's own tendon). Cryoneurolysis is an approved process of applying extreme cold temperatures to targeted nerves in order to decrease or eliminate pain. . If you take part in the research, you will be randomly assigned (assigned by chance, like a flip of a coin) to Group A (standard care) or Group B (standard care plus Cryoneurolysis). Participants in both groups will undergo standard ACL reconstruction and receive standard preoperative and postoperative pain management. Participants in Group B only will also receive a standard treatment of Cryoneurolysis to their surgical knee within 7-10 days before their scheduled surgery. Participants in both groups (A & B) will be asked to bring their remaining postoperative pain medication to their postoperative follow-up appointments for review by study personnel. Participants will also be asked to complete a survey about their knee activity, function and symptoms at these appointments. Your time in the study will last until the completion of the 12-week postoperative follow-up appointment.

ELIGIBILITY:
Inclusion Criteria:

* - Patients aged 14 and over
* Patients who are patients within the PI's practice
* Patients who can speak and read English
* Patients undergoing autograft ACL reconstruction.
* Patients who are opioid naïve

Exclusion Criteria:

* - Under the age of 14
* Non-English speaking/reading patients
* Patients with Reynauds' syndrome
* Patients with skin disorders or hypo-vascularity
* Patients undergoing allograft ACL reconstruction.
* Patients who consistently use opioids preoperatively

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Post-operative opioid consumption | Measured at 1-week, 6-weeks, 12-weeks
  average daily morphine milliequivalents (MMEs) over the measured postoperative period

SECONDARY OUTCOMES:
IKDC Subjective Knee Evaluation Form | 1-week, 6-week, 12-week postoperative period
  10-item self-rated scale measuring symptoms, athletic activity, and knee function.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Virtua Orthopedics Burlington, Burlington, New Jersey
  - Virtua Orthopedics Cherry Hill, Cherry Hill, New Jersey

IPD SHARING:
Plan to Share IPD: No
Will share aggregate data only

REFERENCES:
- [Background] Lung BE, Karasavvidis T, Sharma AK, Amirhekmat A, Stepanyan H, McMaster W, Yang S, So DH. Cryoneurolysis Is a Safe, Effective Modality to Improve Rehabilitation after Total Knee Arthroplasty. Life (Basel). 2022 Aug 29;12(9):1344. doi: 10.3390/life12091344. PMID 36143381
- [Background] Kapadia BH, Berg RA, Daley JA, Fritz J, Bhave A, Mont MA. Periprosthetic joint infection. Lancet. 2016 Jan 23;387(10016):386-394. doi: 10.1016/S0140-6736(14)61798-0. Epub 2015 Jun 28. PMID 26135702
- [Background] Ilfeld BM, Preciado J, Trescot AM. Novel cryoneurolysis device for the treatment of sensory and motor peripheral nerves. Expert Rev Med Devices. 2016 Aug;13(8):713-25. doi: 10.1080/17434440.2016.1204229. Epub 2016 Jul 13. PMID 27333989
- [Background] Dasa V, Lensing G, Parsons M, Harris J, Volaufova J, Bliss R. Percutaneous freezing of sensory nerves prior to total knee arthroplasty. Knee. 2016 Jun;23(3):523-8. doi: 10.1016/j.knee.2016.01.011. Epub 2016 Feb 10. PMID 26875052
- [Result] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454
- [Result] Mihalko WM, Kerkhof AL, Ford MC, Crockarell JR Jr, Harkess JW, Guyton JL. Cryoneurolysis before Total Knee Arthroplasty in Patients With Severe Osteoarthritis for Reduction of Postoperative Pain and Opioid Use in a Single-Center Randomized Controlled Trial. J Arthroplasty. 2021 May;36(5):1590-1598. doi: 10.1016/j.arth.2020.11.013. Epub 2020 Nov 14. PMID 33279353